CLINICAL TRIAL: NCT03841773
Title: A Phase 3, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TNX-102 SL in Participants With PTSD Taken Daily at Bedtime (Protocol No. TNX-CY-P302)
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of TNX-102 SL in Participants With PTSD
Acronym: RECOVERY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim Analysis results
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-P302
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: PTSD
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNX-102 SL Tablet 2.8 mg (Experimental): 2 x TNX-102 SL, 2.8 mg Tablets taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: TNX-102 SL
- Placebo SL Tablet (Placebo Comparator): 2 x Placebo Tablets taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: Placebo SL Tablets

INTERVENTIONS:
Drug: TNX-102 SL — Patients will take 2 tablets of randomly assigned study drug sublingually starting on Day 1 for 12 weeks
  Other Names: Low dose cyclobenzaprine sublingual tablets; Tonmya(R)
  Arms: TNX-102 SL Tablet 2.8 mg
Drug: Placebo SL Tablets — Patients will take 2 tablets of randomly assigned study drug sublingually starting on Day 1 for 12 weeks
  Other Names: Placebo sublingual tablets; TNX-102 SL Placebo Tablets
  Arms: Placebo SL Tablet

SUMMARY:
This is a 12-week, multicenter, randomized, double-blind, placebo-controlled, fixed-dose study that will investigate the efficacy and safety of TNX-102 SL 5.6 mg (2 x 2.8 mg tablets) - a sublingual formulation of cyclobenzaprine. Following successful screening and randomization, eligible patients will have a telephonic visit at week 2 and then return regularly to the study clinic for monthly visits for assessments of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects between the years of 18-75 with a diagnosis of PTSD (diagnosis can be made at screening)
* Index trauma must have occurred within 9 years of Screening Visit
* Must have occurred when the patient was ≥18 years of age

Exclusion Criteria:

* Use of antidepressant medication within 2 months of Baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Sullivan, MD, Study Director — Tonix Pharmaceuticals
Locations (30):
- United States (30):
  - Ashild Peters, Phoenix, Arizona
  - Ashild Peters, Little Rock, Arkansas
  - Ashild Peters, Rogers, Arkansas
  - Ashild Peters, Beverly Hills, California
  - Ashild Peters, Oceanside, California
  - Ashild Peters, Orange, California
  - Ashild Peters, Panorama City, California
  - Ashild Peters, Riverside, California
  - Ashild Peters, San Diego, California
  - Ashild Peters, Temecula, California
  - Ashild Peters, Colorado Springs, Colorado
  - Ashild Peters, Norwich, Connecticut
  - Ashild Peters, Washington D.C., District of Columbia
  - Ashild Peters, Jacksonville, Florida
  - Ashild Peters, North Miami, Florida
  - Ashild Peters, Orlando, Florida
  - Ashild Peters, Tampa, Florida
  - Ashild Peters, Alpharetta, Georgia
  - Ashild Peters, Lincolnwood, Illinois
  - Ashild Peters, Boston, Massachusetts
  - Ashild Peters, New Bedford, Massachusetts
  - Ashild Peters, Flowood, Mississippi
  - Ashild Peters, St Louis, Missouri
  - Ashild Peters, Las Vegas, Nevada
  - Ashild Peters, Oklahoma City, Oklahoma
  - Ashild Peters, Portland, Oregon
  - Ashild Peters, Salem, Oregon
  - Ashild Peters, Memphis, Tennessee
  - Ashild Peters, Austin, Texas
  - Ashild Peters, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- TNX-102 SL Tablet, 5.6 mg: 2 x TNX-102 SL, 2.8 mg Tablets taken sublingually each day at bedtime for 12 weeks.
  TNX-102 SL: Patients will take 2 tablets of randomly assigned study drug sublingually starting on Day 1 for 12 weeks
Period: Overall Study
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 5.6 mg
Started | 93 | 99
Completed | 64 | 59
Not Completed | 29 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 5.6 mg | Total
Number analyzed (Participants) | 93 | 99 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (10.67) | 39.8 (11.61) | 38.5 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 78 | 152
  Male | 19 | 21 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 19 | 35
  Not Hispanic or Latino | 77 | 80 | 157
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 5 | 1 | 6
  Black or African American | 11 | 15 | 26
  White | 71 | 73 | 144
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 93 | 99 | 192

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Total CAPS-5 Score
Description: The primary efficacy endpoint is the mean change from baseline (Day 1) in the total CAPS-5 score after 12 weeks of treatment. The CAPS-5 is an updated and validated version of a semi-structured interview that has been designed to assess the essential features of PTSD as defined by the DSM-5. The total score ranges from 0 to 80 with higher scores indicating more severe PTSD symptoms.
Time Frame: Day 1, Week 12
Population: Results are reported for the mITT population, which includes all randomized participants who have at least a baseline and one post-baseline CAPS-5 assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 5.6 mg
Number analyzed (Participants) | 83 | 80
units on a scale | -18.5 (1.90) | -20.7 (1.97)

2. Secondary Outcome: Clinical Global Impression of Severity (CGI-S)
Description: Change from baseline (Day 1) in CGI-S score at Week 12. CGI-S range from 1 (Normal, not ill at all) to 7 (Among the most extremely ill patients).
Time Frame: Day 1, Week 12
Population: Results are reported for the mITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 5.6 mg
Number analyzed (Participants) | 83 | 80
units on a scale | -1.5 (0.17) | -2.0 (0.18)

3. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: Change from baseline in Sheehan Disability Scale (SDS) total score after 12 weeks of treatment comparing the 5.6 mg treatment arm to placebo. The SDS is a self-report questionnaire that was designed to assess the participant's view of the degree to which symptoms have disrupted work/school, social life/leisure activities, and family life/home responsibilities during the previous two weeks. Score ranges from 0 to 30. A score of 0 means the patient is unimpaired, and a score of 30 means the patient is highly impaired.
Time Frame: Day 1, Week 12
Population: Results are reported for the mITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 5.6 mg
Number analyzed (Participants) | 83 | 80
units on a scale | -7.6 (0.97) | -9.4 (1.01)

4. Secondary Outcome: Patient-Reported Outcome Measurement Information System (PROMIS) Sleep Disturbance
Description: Change from baseline (Day 1) to Week 12 in the PROMIS Sleep Disturbance scale. The PROMIS Sleep disturbance short form 8a consists of 8 questions on a 5-point scale (1 to 5) where a higher score indicates a worse outcome. The total score is reported on a range of 8 to 40. Raw scores are converted to T-scores based on US population with score of 50 as average with a standard deviation of 10.
Time Frame: Day 1, Week 12
Population: Results are reported for the mITT population.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 5.6 mg
Number analyzed (Participants) | 83 | 80
T-score | -9.4 (1.51) | -13.0 (1.57)

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Al Cause Mortality is reported for all participants. AEs and SAEs are reported for the Safety population, which includes participants who took at least 1 dose of study drug.
Arm/Group | Placebo SL Tablet | TNX-102 SL Tablet, 5.6 mg
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/99
Serious Adverse Events (participants affected / at risk) | 2/91 | 0/96
Other Adverse Events (participants affected / at risk) | 17/91 | 46/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SL Tablet (N=91) | TNX-102 SL Tablet, 5.6 mg (N=96)
Cholecystic Acute (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Abcess (Infections and infestations) | 1 | 0
Jaw Fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo SL Tablet (N=91) | TNX-102 SL Tablet, 5.6 mg (N=96)
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 | 28
Dry Mouth (Gastrointestinal disorders) | 3 | 8
Paraesthesia Oral (Gastrointestinal disorders) | 1 | 7
Nausea (Gastrointestinal disorders) | 5 | 1
Tongue Discomfort (Gastrointestinal disorders) | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 5
Headache (Nervous system disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all investigators.

DOCUMENTS (2):
  • Study Protocol (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT03841773/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT03841773/SAP_001.pdf